CLINICAL TRIAL: NCT01795066
Title: Endoscopic Ultrasound-guided Fine Needle Biopsy With 25-gauge Biopsy Needles for Solid Pancreatic Masses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4-2012-0856
Record Dates: First submitted 2013-02-12; First posted 2013-02-20 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2015-12

CONDITIONS: Solid Pancreatic Masses
MeSH Terms: interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EUS-FNB with 25-gauge (Experimental)
  Interventions: Device: EUS-FNB with 25-gauge (Echotip ProCore; Cook Endoscopy Inc, Limerick, Ireland)

INTERVENTIONS:
Device: EUS-FNB with 25-gauge (Echotip ProCore; Cook Endoscopy Inc, Limerick, Ireland)
  Other Names: EUS-FNA with the use of Wilson-Cook procore 25-gauge needles (Echotip, Wilson-Cook, Winston Salem, NC, USA)

SUMMARY:
For 12 months after approvement by the University of Yonsei institutional review board, of the 59 patients older than 20 years referred to our medical center for EUS-FNA or FNB, all consecutive pancreatic lesions were evaluated for inclusion in our prospective study. The inclusion criteria for this study were the following: diagnosed or suspected solid pancreatic masses according to clinical evaluation and imaging studies with need of histologic tissue confirmation by EUS-FNA or EUS-FNB. The exclusion criteria were the following: cystic pancreatic lesions, patients haemodynamically unstable or with severe coagulopathy (international normalized ratio [INR] > 1.5 or platelet count < 50,000 cells/cubic millimeter [cmm3]), patients unable to suspend anticoagulant/anti-platelet therapy, pregnancy, inability or refusal to give informed consent, and refusal to participate in the study. Patients undergoing anticoagulant or anti- platelet therapy for non-critical problems discontinued treatment at least 5 days before the endoscopic procedure. Written informed consent was obtained from all patients for the procedures performed and participation in the study, and the study protocol was approved by the University of Yonsei institutional review board. All patients were underwent the procedure under conscious sedation with propofol and midazolam according to the current guidelines.8 After procedure, the patients were monitored for at least six hours in order to immediately detect post-procedural complications and were followed for up to 7 days in order to detect late complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 20 years referred to our medical center for EUS-FNA or FNB with diagnosed or suspected solid pancreatic masses according to clinical evaluation and imaging studies

Exclusion Criteria:

* cystic pancreatic lesions, patients haemodynamically unstable or with severe coagulopathy (international normalized ratio [INR] > 1.5 or platelet count < 50,000 cells/cubic millimeter [cmm3]), patients unable to suspend anticoagulant/anti-platelet therapy, pregnancy, inability or refusal to give informed consent, and refusal to participate in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01-22 (Actual); Study Completion 2015-01-22 (Actual)

PRIMARY OUTCOMES:
accessing the rate for procurement of the histologic core | up to 5 minuites after endoscopic ultrasound-guided fine needle biopsy
  The tissue samples were immediately fixed in formalin. The histologic cassette was processed, embedded in paraffin, and then prepared in hematoxylin and eosin to be evaluated by one pathologist (K.H.K) for the presence of a histologic core. If the histologic core was present, the specimen was graded as optimal or suboptimal. Optimal specimens were those in which the procured material enabled satisfactory assessment of histologic architecture that either did not change the original diagnosis or yielded additional findings. Suboptimal specimens were those in which the quality of the histologic core was unsatisfactory for assessment of histologic architecture. When required, immunohistochemical or special staining was performed for differentiation of morphologically challenging lesions.10

SECONDARY OUTCOMES:
the percentage of cases in which pathologists classified the sample quality as optimal for histological evaluation of 25-gauge biopsy needle | up to 5 minuites after after endoscopic ultrasound-guided fine needle biopsy
  The tissue samples were immediately fixed in formalin. The histologic cassette was processed, embedded in paraffin, and then prepared in hematoxylin and eosin to be evaluated by one pathologist (K.H.K) for the presence of a histologic core. If the histologic core was present, the specimen was graded as optimal or suboptimal. Optimal specimens were those in which the procured material enabled satisfactory assessment of histologic architecture that either did not change the original diagnosis or yielded additional findings. Suboptimal specimens were those in which the quality of the histologic core was unsatisfactory for assessment of histologic architecture. When required, immunohistochemical or special staining was performed for differentiation of morphologically challenging lesions.10

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Gastroenterology, Department of Internal Medicine, Yonsei Institute of Gastroenterology, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Park SW, Chung MJ, Lee SH, Lee HS, Lee HJ, Park JY, Park SW, Song SY, Kim H, Chung JB, Bang S. Prospective Study for Comparison of Endoscopic Ultrasound-Guided Tissue Acquisition Using 25- and 22-Gauge Core Biopsy Needles in Solid Pancreatic Masses. PLoS One. 2016 May 5;11(5):e0154401. doi: 10.1371/journal.pone.0154401. eCollection 2016. PMID 27149404